CLINICAL TRIAL: NCT03607136
Title: Department of Physical Therapy, Tzu Chi University
Brief Title: Early Detection of Disability and Health Promotion for Community-dwelling Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB106-75-A-2
Record Dates: First submitted 2018-07-05; First posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Elderly; Sarcopenia
Keywords: early detection; health promotion; community-dwelling; elderly
MeSH Terms: conditions — Sarcopenia | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise training (Experimental): Participants in the exercise training group received a 12-week exercise training.
  Interventions: Other: exercise training
- control (No Intervention): Participants in the control group did not receive any specific training programs instead of maintaining their usual activities of daily living.

INTERVENTIONS:
Other: exercise training — Aerobic exercises, strengthening exercises, flexibility training for 60min, twice a week for 12 weeks
  Arms: exercise training

SUMMARY:
This study evaluates the effects of exercise intervention on muscle strength and walking speed for the community-dwelling elderly. Half of the participants will receive exercise training, while the other half will maintain their usual activities of daily living.

DETAILED DESCRIPTION:
Physical inactivity can result in physical frailty and sarcopenia. Physical frailty and sarcopenia are two common and mostly overlapping geriatric conditions, which may cause negative consequences of aging, such as disability, hospitalization and mortality.

Regular physical activity has been suggested to maintain or improve functional capacity and body composition, as well as delay aging process. Nevertheless, inactivity prevalence still significantly increases among older adults, especially those with a disability. One of the probable reasons is that the use of physical activities or exercise interventions is not tailored to the needs and capabilities of the elderly.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 50 years
* able to follow simple instructions
* willing to participate and sign consent form

Exclusion Criteria:

* unstable angina or epilepsy
* severe visual deficits
* cognitive dysfunction
* other musculoskeletal conditions that will limit mobility

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Walking speed | Change from baseline at 12 weeks
  Participants are asked to walk along a 14 m hallway. The time taken to the middle 10 m is recorded to calculate walking speed (m/s).
Muscle strength | Change from baseline at 12 weeks
  Muscle strength is assessed using hand-hold Dynamometers

SECONDARY OUTCOMES:
Timed up and go test | Change from baseline at 12 weeks
  Participants are asked to stand up, walk 3 m, turn around a cone, and return to a sitting position
Walking endurance | Change from baseline at 12 weeks
  Participants are asked to walk back and forth along a 20-meter corridor and to cover the maximum distance possible in six minutes
Sit-to-stand test | Change from baseline at 12 weeks
  Participants are asked to stand up and sit down 5 times.
Berg balance scale | Change from baseline at 12 weeks
  It consists of 14 items, including sitting unsupported, standing unsupported, standing with eyes closed, standing with feet together, standing on one foot, turning to look behind, retrieving objective from floor, random standing, reaching forward with an outsrptretched arm, sit to stand, stand to sit, transfer, turning 360 degrees, stool stepping, scored from 0 to 4, "0" indicates the lowest level of function and "4" the highest level of function. Total Score = 56.
Gait kinematics | Change from baseline at 12 weeks
  Gait kinematics are assessed by angular displacement of lower limbs using shoe-worn inertial measurement unit based device